CLINICAL TRIAL: NCT02385682
Title: CardiOvascular Risk and idEntificAtion of Potential High-risk Population in Korean Patients With Acute Myocardial Infarction Registry (COREA-AMI)
Brief Title: CardiOvascular Risk and idEntificAtion of Potential High-risk Population in Acute Myocardial Infarction
Acronym: COREA-AMI
Status: Completed | Type: Observational
Sponsor: Kiyuk Chang (Other)
Collaborators: The Catholic University of Korea (Other); Chonnam National University (Other)
Responsible Party: Sponsor-Investigator, Kiyuk Chang, Chief of the division of cardiology, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Other Study IDs: XC13RIMI0060k
Record Dates: First submitted 2015-03-05; First posted 2015-03-11 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Long-term Major Cardiovascular Events; Myocardial Infarction; Percutaneous Coronary Intervention
MeSH Terms: conditions — Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ST-segment elevation AMI: ST-segment elevation acute myocardial infarction teated with percutaneous coronary intervention
  Interventions: Device: Percutaneous coronary intervention
- Non-ST-segment elevation AMI: Non-ST-segment elevation acute myocardial infarction teated with percutaneous coronary intervention
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — Percutaneous coronary intervention
  Groups: Non-ST-segment elevation AMI
Device: Percutaneous coronary intervention — Percutaneous coronary intervention
  Groups: ST-segment elevation AMI

SUMMARY:
The purpose of this registry is to evaluate long-term clinical events in patients with acute myocardial infarction who were treated with percutaneous coronary intervention.

Although numerous articles have been published by using nationwide Korean myocardial infarction registries, such as the Korea Acute Myocardial Infarction Registry (KAMIR), limitation of previous registries is that these have little data beyond the first year of MI. Therefore, current registry was designed to assess long-term clinical events in patients with acute myocardial infarction.

Because most of myocardial infarction patients were treated by revascularization in real world of Korea, this registry limits the inclusion criteria to patients who were treated with percutaneous coronary intervention to reduce the bias.

DETAILED DESCRIPTION:
Cardiovascular center with high-volume percutaneous coronary intervention of following hospitals were participated.

* Seoul St. Mary's Hospital, Seoul, South Korea
* Yeoido St. Mary's Hospital, Seoul, South Korea
* Uijongbu St. Mary's Hospital, Gyeonggi-do, South Korea
* St. Paul Hospital, Seoul, South Korea
* Bucheon St. Mary's Hospital, Gyeonggi-do, South Korea
* Incheon St. Mary's Hospital, Incheon, South Korea
* St. Vincent Hospital, Gyeonggi-do, South Korea
* Deajon St. Mary's Hospital, Daejeon, South Korea
* Cheonnam University Hospital, Gwangju, South Korea

  8 hospitals of the Catholic University of Korea already have web-based coronary intervention registry (NCT01239914). And Cheonnam University Hospital is one of leading hospitals to design and manage the web-based previous Korean nationwide myocardial infarction registry, such as such as the Korea Acute Myocardial Infarction Registry (KAMIR) (http://www.kamir.or.kr/).

All consecutive acute myocardial infarction patients had been enrolled in each registries prospectively.

Using these previous data, current registry update new clinical and angiographic variables and assess long-term clinical follow-up data retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction who were treated with percutaneous coronary intervention

Exclusion Criteria:

* Acute myocardial infarction who were managed by conservative strategy
* Acute myocardial infarction who were not treated with percutaneous coronary intervention

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute myocardial infarction who were treated with percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 4748 (Actual)
Dates: Start 2004-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events | 5 years

SECONDARY OUTCOMES:
All-cause death | 5 years
Cardiac death | 5 years
Nonfatal myocardial infarction | 5 years
Nonfatal stroke | 5 years
Target lesion revascularization | 5 years
Target vessel revascularization | 5 years
Non-target vessel revascularization | 5 years
Definite/Probable stent thrombosis | 5 years
Hospitalization for heart failure | 5 years
Bleeding defined as the Bleeding Academic Research Consortium (BARC) definitions type 2, 3, and 5 | 5 years
Bleeding defined as the thrombolysis In Myocardial Infarction (TIMI) major/minor | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Bae Seung, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital; Myung Ho Jeong, MD, PhD, Principal Investigator — Chonnam National University Hospital

REFERENCES:
- [Derived] Ahn Y, Lee D, Choo EH, Choi IJ, Lim S, Lee KY, Hwang BH, Park MW, Lee JM, Park CS, Kim HY, Yoo KD, Jeon DS, Chung WS, Kim MC, Jeong MH, Ahn Y, Chang K. Association Between Bleeding and New Cancer Detection and the Prognosis in Patients With Myocardial Infarction. J Am Heart Assoc. 2022 Nov 15;11(22):e026588. doi: 10.1161/JAHA.122.026588. Epub 2022 Nov 8. PMID 36346059
- [Derived] Lim S, Choo EH, Choi IJ, Ihm SH, Kim HY, Ahn Y, Chang K, Jeong MH, Seung KB. Angiotensin Receptor Blockers as an Alternative to Angiotensin-Converting Enzyme Inhibitors in Patients with Acute Myocardial Infarction Undergoing Percutaneous Coronary Intervention. J Korean Med Sci. 2019 Nov 25;34(45):e289. doi: 10.3346/jkms.2019.34.e289. PMID 31760711
- [Derived] Kim MC, Ahn Y, Cho JY, Lee KH, Sim DS, Yoon NS, Yoon HJ, Kim KH, Hong YJ, Park HW, Kim JH, Jeong MH, Cho JG, Park JC, Chang K, Seung KB. Benefit of Early Statin Initiation within 48 Hours after Admission in Statin-Naive Patients with Acute Myocardial Infarction Undergoing Percutaneous Coronary Intervention. Korean Circ J. 2019 May;49(5):419-433. doi: 10.4070/kcj.2018.0341. Epub 2019 Feb 12. PMID 30808084